CLINICAL TRIAL: NCT01072188
Title: Clinical Efficacy of 10% Arginine Bicarbonate Prophylaxis Paste
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2008-07-SEN-PROPREC-ED
Record Dates: First submitted 2008-09-26; First posted 2010-02-19 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ProClude Prophylaxis paste-A (Active Comparator): Arginine Bicarbonate prophylaxis paste
  Interventions: Device: Arginine/Calcium Carbonate
- Nupro-M Prophylaxis paste -B (Placebo Comparator): Control prophylaxis paste (Fluoride free - placebo)
  Interventions: Device: Nupro - Fluoride Free

INTERVENTIONS:
Device: Arginine/Calcium Carbonate — One time treatment
  Arms: ProClude Prophylaxis paste-A
Device: Nupro - Fluoride Free — Brush twice daily
  Arms: Nupro-M Prophylaxis paste -B

SUMMARY:
The objective of this study is to evaluate the clinical efficacy of a prophylaxis paste containing 10% arginine bicarbonate on dentinal hypersensitivity reduction when applied as a pre-procedure to a professional dental cleaning.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.
* Availability for the three (3) week duration of the study.
* Two (2) sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to tactile stimuli (Yeaple probe) as defined by a score between 10-50gms. of force.
* Qualifying response to the air blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both the parameters assessed (tactile or air) on two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for three months prior to entry into the study.
* Signed Informed Consent Form.

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Scheduled dental prophylaxis within three weeks prior to the Baseline Hypersensitivity Examination.
* Sensitive teeth with mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Subjects that began to take anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily analgesics within one month prior to the start of the study or who have to start taking these during the course of the study.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past three months.
* Current participation in any other clinical study.
* Pregnant or lactating subjects.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hamlin, DDS, Principal Investigator — Contract Dental Evaluations
Locations (1):
- Contract Dental Evaluations, Langhorne, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ProClude Prophylaxis Paste-A: Arginine Bicarbonate prophy paste (experimental).
- Nupro-M Prophylaxis Paste-B: Control prophy paste (Fluoride free).
Period: Overall Study
Arm/Group | ProClude Prophylaxis Paste-A | Nupro-M Prophylaxis Paste-B
Started | 22 | 23
Completed | 22 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProClude Prophylaxis Paste-A | Nupro-M Prophylaxis Paste-B | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 44.13 (7.78) | 45.91 (11.41) | 45 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Hypersensitivity to Touch (Tactile)
Description: Units on a scale: Measured with an electronic force sensing probe (Yeaple Probe): 10, 20, 30, 40, up to 50 grams of force are applied to hypersensitive tooth until pain elicited. Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. The higher the score, the higher the hypersensitivity.
Time Frame: Immediately after product application
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ProClude Prophylaxis Paste-A | Nupro-M Prophylaxis Paste-B
Number analyzed (Participants) | 22 | 23
Units on a scale | 42.2 (9.25) | 20.1 (9.25)
Statistical Analysis 1: Comparison: ProClude Prophylaxis Paste-A vs Nupro-M Prophylaxis Paste-B; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Air Blast
Description: Units on a scale using Schiff Cold Air Sensitivity Scale. Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth. According to this analog scale hypersensitivity scores for the stimulated tooth is 0, 1, 2 or 3(The lower the score, the lower the hypersensitivity). 0=No subject response to stimulus, 1=responds but will continue, 2=responds and moves or requests discontinuation, 3=Painful response to stimulus, discontinuation requested.
Time Frame: Immediately after product application
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ProClude Prophylaxis Paste-A | Nupro-M Prophylaxis Paste-B
Number analyzed (Participants) | 22 | 23
Units on a scale | 1.26 (0.58) | 2.17 (0.58)
Statistical Analysis 1: Comparison: ProClude Prophylaxis Paste-A vs Nupro-M Prophylaxis Paste-B; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | ProClude Prophylaxis Paste-A | Nupro-M Prophylaxis Paste-B
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days